CLINICAL TRIAL: NCT06926647
Title: A Multicenter, Prospective, Real-World Study of Antiviral Therapy in Children With Chronic Hepatitis B
Brief Title: A Real-World Study of Antiviral Therapy in Children With Chronic Hepatitis B
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Chief physician, Beijing 302 Hospital
Other Study IDs: KY-2025-2-31-2
Record Dates: First submitted 2025-04-11; First posted 2025-04-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: HBV; Chronic Hepatitis b
Keywords: Nucleos(t)ide Analogues（NAs）; Interferon alpha（IFNα）
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Interferon-alpha

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Initial Treatment Cohort 1
  Interventions: Drug: Nucleos(t)ide Analogues; Drug: Interferon alfa; Drug: NAs combined with IFNα; Other: comparative observation
- Previously Treated Cohort 1
  Interventions: Drug: Nucleos(t)ide Analogues; Drug: NAs combined with IFNα; Other: drug withdrawal observation

INTERVENTIONS:
Drug: Nucleos(t)ide Analogues — Administer NAs [LAM, ETV, TDF, TAF (TAF preferred for those aged 6 years and older)] continuously for 48 weeks based on age.
Drug: Interferon alfa — IFNα monotherapy for 48 weeks (select conventional IFNα for ages ≥1 and <3 years, select PEG-IFNα-2b for ages ≥3 years)
  Groups: Initial Treatment Cohort 1
Drug: NAs combined with IFNα — Receive NAs combined with IFNα treatment for 48 weeks.
Other: comparative observation — Blank control observation for 48 weeks.
  Groups: Initial Treatment Cohort 1
Other: drug withdrawal observation — This group is the drug withdrawal observation group, which will strictly monitor virological indicators and biochemical results, and will reinitiate antiviral treatment if necessary based on antiviral treatment standards and the willingness of the child (or family members)
  Groups: Previously Treated Cohort 1

SUMMARY:
This is a multicenter, prospective, real-world study. The study plans to include a total of 2000 patients who meet the inclusion and exclusion criteria, consisting of 1600 treatment-naive patients and 400 treatment-experienced patients. The effectiveness and safety of different treatment strategies will be evaluated in children aged 1-12 years with treatment-naive and treatment-experienced chronic hepatitis B (CHB) and chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Initial Treatment Group:

  1. The guardian understands and signs the informed consent form (both parents must sign), and adheres to the relevant requirements of this study. If the participant is 8 years old or older, they must also sign the informed consent form. For participants under 8 years old who can express consent, their consent must be clearly documented.
  2. Age: ≥1 year and <13 years, either sex;
  3. Positive for HBsAg and/or HBV DNA for more than 6 months;
  4. No prior antiviral treatment.
* Treated Group:

  1. The guardian understands and signs the informed consent form (both parents must sign), and adheres to the relevant requirements of this study. If the participant is 8 years old or older, they must also sign the informed consent form. For participants under 8 years old who can express consent, their consent must be clearly documented.
  2. Age: ≥3 years and <13 years, either sex;
  3. Previously diagnosed with chronic hepatitis B and received antiviral treatment with NAs for more than 1 year and currently on treatment;
  4. No history of IFNα use in the past 6 months;
  5. Negative for HBV DNA;
  6. HBsAg quantification <10,000 IU/ml (HBsAg can be negative in the drug discontinuation observation group);
  7. The drug discontinuation observation group must also achieve negative HBV DNA and HBeAg seroconversion for at least 1 year (based on continuous results from three consecutive reviews), and HBsAg <10,000 IU/ml; NAs will be discontinued after enrollment.

Exclusion Criteria:

* 1.In the interferon group, blood white blood cell count <3.5×10^9/L, or platelet count <80×10^9/L, or prothrombin activity <60%, or total bilirubin >34μmol/L, or serum albumin <35g/L, or serum creatinine >133μmol/L; 2.Coexistence of other active infections; 3. Coexistence of other chronic liver diseases or active liver diseases, such as autoimmune liver disease, drug-induced liver injury, Wilson's disease, decompensated cirrhosis, liver cancer; 4. Coexistence of other severe systemic diseases or malignant tumors, etc.; 5. History of allergy to nucleoside analogues or interferon; 6. Subjects whom the investigator deems to have poor compliance, unable or unwilling to provide informed consent, or unable to adhere to the study requirements, or other conditions not suitable for participation in this study.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients provided by hospitals from various centers across the country are standardized in English translation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg seroconversion rate | Week 48,96

SECONDARY OUTCOMES:
HBV DNA negative conversion rate | Week 48,96
HBeAg negative conversion rate | Week 48,96
HBeAg seroconversion rate | Week 48,96
HBsAg seroconversion rate | Week 48,96
ALT normalization rate | Week 48,96

CONTACTS AND LOCATIONS:
Overall Officials: Fusheng Wang, Study Director — Fifth Medical Center of Chinese PLA General Hospital
Locations (84):
- China (84):
  - Ankang Central Hospital, Ankang
  - Anyang Fifth People's Hospital, Anyang
  - Beihai People's Hospital, Beihai
  - 301 Hospital, Beijing
  - Binzhou Medical University Affiliated Hospital, Binzhou
  - Changzhi Medical College Affiliated Peace Hospital, Changzhi
  - Changzhou Third People's Hospital, Changzhou
  - Chengdu Public Health Clinical Medical Center, Chengdu
  - West China Second Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Dongguan People's Hospital, Dongguan
  - Dongying People's Hospital, Dongying
  - Foshan First People's Hospital, Foshan
  - Southern Medical University Shunde Hospital, Foshan
  - Guangzhou Medical University Affiliated Women and Children's Medical Center, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Hainan Women and Children's Medical Center, Haikou
  - Handan Infectious Disease Hospital, Handan
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Hepu County People's Hospital, Hepu
  - Shanxian Central Hospital, Heze
  - Jiangmen Traditional Chinese Medicine Hospital, Jiangmen
  - Lanzhou Second People's Hospital, Lanzhou
  - Tibet Autonomous Region Third People's Hospital, Lhasa
  - Liaocheng People's Hospital, Liaocheng
  - Linfen People's Hospital, Linfen
  - Linfen Third People's Hospital, Linfen
  - Liuzhou Workers' Hospital, Liuchow
  - Longyan Second Hospital, Longyan
  - Luoyang Central Hospital, Luoyang
  - Southwest Medical University Affiliated Hospital, Luzhou
  - Jiangxi Children's Hospital, Nanchang
  - Nanchang Ninth Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanning Fourth People's Hospital, Nanning
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nanyang Central Hospital, Nanyang
  - Affiliated Hospital of Putian University, Putian
  - Putian First Hospital, Putian
  - Qingdao Public Health Clinical Center, Qingdao
  - Quanzhou Maternal and Child Health Hospital Children's Hospital, Quanzhou
  - Queshan County People's Hospital, Queshan
  - Shangcheng County People's Hospital, Shangcheng
  - Shanghai Children's Hospital, Shanghai
  - Shangqiu City Hospital, Shangqiu
  - Shangqiu First People's Hospital, Shangqiu
  - Shangqiu Third People's Hospital, Shangqiu
  - Northern Guangdong Second People's Hospital, Shaoguan
  - Shenzhen Third People's Hospital, Shenzhen
  - The First Affiliated Hospital of Shihezi University, Shihezi
  - Handan Infectious Disease Hospital, Shijiazhuang
  - Shijiazhuang Fifth Hospital, Shijiazhuang
  - Suzhou Fifth People's Hospital, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - Taiyuan Third People's Hospital, Taiyuan
  - Taian Central Hospital, Tai’an
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Xinjiang Uygur Autonomous Region Infectious Diseases Hospital, Ürümqi
  - Weifang Medical University Affiliated Hospital, Weifang
  - Weishi County People's Hospital, Weishi
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Air Force Medical University (Tangdu Hospital), Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Traditional Chinese Medicine Hospital, Xiamen
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen
  - Liangshan Yi Autonomous Prefecture Seventh People's Hospital, Xichang
  - Qinghai Fourth People's Hospital, Xining
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Xixian People's Hospital, Xixian
  - Xuchang Central Hospital, Xuchang
  - Xuchang People's Hospital, Xuchang
  - Yantai Qishan Hospital, Yantai
  - Yongcheng People's Hospital, Yongcheng
  - Yulin Traditional Chinese Medicine Hospital, Yulin
  - Yuncheng Central Hospital, Yuncheng
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou
  - Zhongshan Second People's Hospital, Zhongshan
  - Zhumadian Central Hospital, Zhumadian
  - Zibo Infectious Diseases Hospital, Zibo

IPD SHARING:
Plan to Share IPD: No